CLINICAL TRIAL: NCT00812409
Title: Resistance and Aerobic Exercise With Nutritional Supplementation in Men and Women
Acronym: S-017
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Wayne Campbell, Ph.D., Purdue University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0611004694; 07053552
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Obesity
Keywords: Measuring markers of metabolic syndrome in overweight and obese adults.
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): Control group: non-protein supplement with resistance and aerobic exercise.
  Interventions: Other: Non protein supplementation with exercise (control)
- 2 (Experimental): Low protein supplement with resistance and aerobic exercise.
  Interventions: Dietary Supplement: Whey protein supplementation with exercise
- 3 (Experimental): Moderate protein supplement with resistance and aerobic exercise.
  Interventions: Dietary Supplement: Whey protein supplementation with exercise
- 4 (Experimental): High protein supplement with resistance and aerobic exercise.
  Interventions: Dietary Supplement: Whey protein supplementation with exercise

INTERVENTIONS:
Dietary Supplement: Whey protein supplementation with exercise — Whey protein supplementation with resistance and aerobic exercise.
  Arms: 2; 3; 4
Other: Non protein supplementation with exercise (control) — Non protein supplementation with resistance and aerobic exercise.
  Arms: 1

SUMMARY:
The purpose of this study is to identify the influence of resistance and aerobic exercise with different nutritional supplements in middle-aged men and women on various physiological measures. Throughout the study, the investigators examine body composition, body weight, food intake, fitness level, metabolism, and blood hormones.

ELIGIBILITY:
Inclusion Criteria:

* men and women age 35-65 yr
* body weight <300 lbs (136 kg)
* body mass index between 28 kg/m2 and 35 kg/m2
* fasting glucose <110 mg/dL
* blood pressure <160/100 mm Hg
* plasma total cholesterol <260 mg/dL
* LDL-cholesterol <160 mg/dL
* triacylglycerol <400 mg/dL
* not currently or previously following a weight loss diet or other special/non-balanced diet (in the past 6 months)
* <1 hour/week of habitual aerobic exercise training and no resistance
* exercise training (in the past 6 months)

Exclusion Criteria:

* men and women age < 35 yr or >65 yr
* body weight >300 lbs (136 kg)
* body mass index between <28 kg/m2 or >35 kg/m2
* fasting glucose >110 mg/dL
* blood pressure >160/100 mm Hg
* plasma total cholesterol >260 mg/dL
* LDL-cholesterol >160 mg/dL
* triacylglycerol >400 mg/dL
* currently or previously following a weight loss diet or other special/non- balanced diet (in the past 6 months)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2007-04; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Influence of resistance and aerobic exercise and whey protein on body weight and body composition (fat mass and fat free mass). | 36 weeks

SECONDARY OUTCOMES:
Influence of resistance and aerobic exercise and whey protein on dietary and macronutrient intakes, insulin-mediated glucose metabolism, physical fitness and markers of metabolic and cardiovascular health. | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, Ph.D., Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Wright CS, McMorrow AM, Weinheimer-Haus EM, Campbell WW. Whey Protein Supplementation and Higher Total Protein Intake Do Not Influence Bone Quantity in Overweight and Obese Adults Following a 36-Week Exercise and Diet Intervention. J Nutr. 2017 Feb;147(2):179-186. doi: 10.3945/jn.116.240473. Epub 2016 Dec 21. PMID 28003538
- [Derived] Wright CS, Weinheimer-Haus EM, Fleet JC, Peacock M, Campbell WW. The Apparent Relation between Plasma 25-Hydroxyvitamin D and Insulin Resistance is Largely Attributable to Central Adiposity in Overweight and Obese Adults. J Nutr. 2015 Dec;145(12):2683-9. doi: 10.3945/jn.115.220541. Epub 2015 Oct 7. PMID 26446485
- [Derived] Campbell WW, Kim JE, Amankwaah AF, Gordon SL, Weinheimer-Haus EM. Higher Total Protein Intake and Change in Total Protein Intake Affect Body Composition but Not Metabolic Syndrome Indexes in Middle-Aged Overweight and Obese Adults Who Perform Resistance and Aerobic Exercise for 36 Weeks. J Nutr. 2015 Sep;145(9):2076-83. doi: 10.3945/jn.115.213595. Epub 2015 Aug 5. PMID 26246322
- [Derived] Weinheimer EM, Conley TB, Kobza VM, Sands LP, Lim E, Janle EM, Campbell WW. Whey protein supplementation does not affect exercise training-induced changes in body composition and indices of metabolic syndrome in middle-aged overweight and obese adults. J Nutr. 2012 Aug;142(8):1532-9. doi: 10.3945/jn.111.153619. Epub 2012 Jun 20. PMID 22718030